CLINICAL TRIAL: NCT06061406
Title: BE Smart - Bariatric Patient - Empowerment in the Preparation and Follow-up of Bariatric Surgery Using the Smartvisit App (BESmart)
Acronym: BESmart
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: aycan Medical Systems LTD, Innere Aumuehlstr. 5, 97076 Wuerzburg , Germany (Unknown)
Responsible Party: Principal Investigator, Ann-Cathrin Koschker, Head of outpatient clinic for diabetes and lipids, Wuerzburg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BESmart 228/20
Record Dates: First submitted 2022-03-31; First posted 2023-09-29 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: App; Empowerment; Obesity; bariatric surgery
MeSH Terms: conditions — Obesity; Alzheimer Disease; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group1 (Experimental): Bariatric-metabolic surgery (Gastric sleeve, Roux-Y gastric bypass, omega-loop bypass) at least 24 months ago, 25-45 patients in this group (total sum of patients in all three groups: 100).
  Interventions: Device: smart visit app
- group 2 (Experimental): Patients participating in a full or partial (if primary indication) multimodal approach prior to bariatric surgery, 25-45 patients in this group (total sum of patients in all three groups: 100).
  Interventions: Device: smart visit app
- group 3 (Experimental): Conservative therapy: patients with overweight/obesity grade 1 (BMI 28-34.9 kg/m2), 25-45 patients in this group (total sum of patients in all three groups: 100).
  Interventions: Device: smart visit app

INTERVENTIONS:
Device: smart visit app — Patients use an obesity-adapted version of aycan's Smartvisit app, which helps track specific behaviors (diet, exercise), query potential problems/complaints, and manage medical documents in a structured way.
  A study nurse experienced in the field of nutrition/obesity contacts the patient if necessary and establishes contact with the center physician.

SUMMARY:
Obesity affects an increasing proportion of the population and is associated with numerous comorbidities that cause increased morbidity and mortality.

The most effective therapy for morbid obesity is metabolic bariatric surgery. Surgical numbers are increasing worldwide. Before surgery, patients must try to reduce weight conservatively in a multimodal therapy concept. In addition, numerous protocols must be collected and appointments must be organized. Postoperatively, patients are expected to receive lifelong follow-up care, which increasingly overwhelms bariatric centers.

People with overweight and obesity ° I are often left largely alone with the treatment of their disease. There is a considerable gap in care here.

For the care of patients with obesity and empowerment in dealing with their disease, the smart visit app from the company aycan, which is adapted to obesity patients, is to be investigated. This is designed as a pilot project with the primary endpoint of usage and satisfaction (after 3 months, key secondary endpoint after 12 months). A total of 100 patients from 3 groups (postoperative, preoperative, permanent conservative with only overweight/obesity °I) will use the app for 1 year for this purpose.

DETAILED DESCRIPTION:
The prevalence of obesity has been increasing dramatically for decades. The comorbidities are manifold, and the treatment of obesity is a long-term, usually lifelong task. Metabolic-bariatric surgery offers the best results. However, even after bariatric-metabolic surgery, there is a need for lifelong follow-up to ensure the success of therapy and to identify and treat possible complications, nutritional problems or deficiencies in a timely manner.

The treating centers are increasingly overwhelmed by the follow-up care of the numerous patients. At the same time, the guidelines of the professional societies recommend involving the patient in the success of his or her therapy and enabling him or her to play an active role in shaping his or her treatment. An app tailored to the treatment of obese people, which helps both in the self-organization of the patients in complying with the therapy recommendations and in maintaining contact with the center on a permanent basis and making low-threshold contact when necessary, would be a valuable addition to the existing therapy options for patients and centers alike.

Such an app would also have its value in the preoperative patient, especially since a lot of documentation work has to be done by the patient in this phase.

Patients whose obesity is not pronounced enough for a surgical procedure often complete nutritional counseling and exercise at their own expense without receiving support from experts. Here, too, there would be a need to supplement the therapy options with an appropriately coordinated app.

For the care of patients with obesity and empowerment in dealing with their disease, the smart visit app from the company aycan, which is adapted to obesity patients, is to be investigated. This is designed as a pilot project with the primary endpoint of usage and satisfaction (after 3 months, key secondary endpoint after 12 months). A total of 100 patients from 3 groups (postoperative, preoperative, permanent conservative with only overweight/obesity °I) will use the app for 1 year for this purpose.

ELIGIBILITY:
General inclusion criteria:

* Smartphone available (iOS or Android with sufficient version of the operating system).
* Age >/= 18 years
* Sufficient language skills to answer the questionnaires

Additional group specific inclusion criteria:

Group 1 (bariatric-metabolic surgery):

• Bariatric-metabolic surgery (sleeve gastrectomy, Roux-Y gastric bypass, omega-loop bypass) at least 24 months ago.

Group 2 (multimodal treatment):

• Participation in a full or partial (if primary indication) multimodal approach.

Group 3 (conservative therapy):

* BMI 28-34.9 kg/m2
* No planned bariatric-metabolic surgery
* Desire for conservative weight reduction

Exclusion Criteria:

• current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
satisfaction with and use of smart visit app designed for obesity them self-manage their condition. Analysis of all 3 groups cumulated. Coprimary endpoint | at 3 months
  acceptance: questionnaire assessing the satisfaction with the app (scale 0-100, 0 meaning least possible satisfaction, 100 meaning best possible satisfaction) use: precentage of entered values in the app of the intended values (scale 0-100, 0 meaning no entered values, 100 meaning all intented values were entered)

SECONDARY OUTCOMES:
satisfaction with and use of smart visit app designed for obesity them self-manage their condition. Analysis of all 3 groups cumulated. Coprimary endpoint. | at 12 months
  acceptance: questionnaire assessing the satisfaction with the app (scale 0-100, 0 meaning least possible satisfaction, 100 meaning best possible satisfaction) use: precentage of entered values in the app of the intended values (scale 0-100, 0 meaning no entered values, 100 meaning all intented values were entered)
change in weight | at 3 months and 12 months
  change in weight in kilograms
change in quality of life by SF-36 | at 3 months and 12 months
  measured by SF-36 (short form-36) questionnaire, z-transformed scale, 0 meaning worst possible quality of life, 100 meaning best possible quality of life
change in obesity related quality of life by BQL | at 3 months and 12 months
  measured by BQL (bariatric quality of life) questionnaire index, 0 meaning worst possible quality of life, 100 meaning best possible quality of life
change in quality of life by EQ-5D-5L | at 3 months and 12 months
  measured by EQ-5D-5L questionnaire (European Quality of Life 5 Dimensions 5 Level Version)
Depressive symptoms | at 3 months and 12 months
  measured by PHQ-9 questionnaire (Public Health Questionnaire-9), 0 meaning least possible depressive symptoms, 27 meaning worst possible depressive symptoms
Eating behavior | at 3 months and 12 months
  measured by EDE-Q8 (Eating Disorder Examination Questionnaire Short Version)
Number of contacts patient - center via app | at 3 months and 12 months
  Number of contacts between patients and center via app
daily step counts | at 3 months and 12 months
  change in daily step counts as measured with a pedometer
daily protein intake | at 3 months and 12 months
  change in daily protein intake (entered into the app) in grams
daily calory intake | at 3 months and 12 months
  change in daily calory intake (entered into the app) in kcal
walking distance in 6 minute walk test | at 3 months and 12 months
  change in walking distance in the 6 minute walk test in meters
body composition: body fat measured by bioelectrical impedance analysis | at 3 months and 12 months
  change in body fat (in %)
body composition: phase angle measured by by bioelectrical impedance analysis | at 3 months and 12 months
  change in phase angle (in °)
vitamin B 12 deficiency (only group 1) | at 3 months and 12 months
  vitamin B12 levels below the lower limit of normal
folic acid deficiency (only group 1) | at 3 months and 12 months
  folic acid levels below the lower limit of normal, ferritin, hemoglobin, prealbumin, 25-OH vitamin D, zinc (only group 1)
iron deficiency (only group 1) | at 3 months and 12 months
  ferritin below the lower limit of normal
protein malnutrition (only group 1) | at 3 months and 12 months
  prealbumin below the lower limit of normal
vitamin D deficiency (only group 1) | at 3 months and 12 months
  25-OH vitamin D below the lower limit of normal
zinc deficiency (only group 1) | at 3 months and 12 months
  zinc below the lower limit of normal

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrin D Koschker, Principal Investigator — University Hospital Wuerzburg
Locations (1):
- Ann-Cathrin D Koschker, Würzburg, Germany